CLINICAL TRIAL: NCT06947213
Title: Fragile Bones, Strong Obsessions: A Controlled Study on Orthorexia Nervosa, Body Image and Mood in Postmenopausal Women With Osteoporosis
Brief Title: Orthorexia Nervosa in Postmenopausal Osteoporosis
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: Beylikdüzüstateh17
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A total of 64 female patients diagnosed with osteoporosis based on dual-energy X-ray absorptiometry (DXA) measurements performed within the last six months, and 64 age-matched healthy controls without osteoporosis, will be included in our study. Sociodemographic data such as age, sex, height, weight, and BMI will be recorded. Additionally, information regarding the duration of osteoporosis diagnosis, current treatments, history of fractures, history of falls, comorbidities, and smoking status will be collected. Femoral neck and L1-L4 T-scores and bone mineral density values obtained from existing DXA scans will be documented. Orthorexia nervosa-related symptoms will be assessed using the ORTO-11 scale, mood will be evaluated using the Hospital Anxiety and Depression Scale (HADS), and body image will be assessed using the Body Appreciation Scale-2.

ELIGIBILITY:
Inclusion Criteria:

* Women between 55-75 years
* Women diagnosed with osteoporosis based on DXA measurements performed within the past six months.
* Women aged similarly to the osteoporosis group without a diagnosis of osteoporosis (healthy controls).
* Willingness to participate and provision of written informed consent.

Exclusion Criteria:

* Refusal to participate in the study.
* Diagnosed psychiatric disorders.
* Cognitive impairment.
* Presence of malignancy.
* Presence of endocrine disorders (e.g., hyperthyroidism, Cushing's syndrome).
* Use of glucocorticoids.
* Use of medications affecting mood.

Ages: 55 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study population will consist of postmenopausal women with osteoporosis and age-matched healthy controls
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
ORTO-11 Scale | Baseline
  The ORTO-11 assesses orthorexic tendencies, which refer to an unhealthy obsession with healthy eating. It consists of 11 items rated on a 4-point Likert scale. Total scores range from 11 to 44, with lower scores indicating a higher risk of orthorexia nervosa.

SECONDARY OUTCOMES:
Body Appreciation Scale-2 (BAS-2) | Baseline
  The BAS-2 assesses positive body image and appreciation of one's body. It consists of 10 items rated on a 5-point Likert scale (1 = Never, 5 = Always). Total scores range from 10 to 50, with higher scores indicating greater body appreciation.

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale (HADS)- Anxiety Score | Baseline
  The HADS-A subscale evaluates symptoms of anxiety. It consists of 7 items, each scored between 0 and 3. The total score ranges from 0 to 21, with higher scores indicating higher levels of anxiety.
Hospital Anxiety and Depression Scale (HADS)- Depression Score | Baseline
  The HADS-D subscale evaluates symptoms of depression. It consists of 7 items, each scored between 0 and 3. The total score ranges from 0 to 21, with higher scores indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Turkey (Türkiye)